CLINICAL TRIAL: NCT04772963
Title: Genetics of Central Nervous System Arteriovenous Malformations (AVM): Genotype-Phenotype Correlation and Prognostic Impact on Patients With AVM
Brief Title: Genetics of Central Nervous System Arteriovenous Malformations (GENE-MAV)
Acronym: GENE-MAV
Status: Recruiting | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: SSA_2021_3
Record Dates: First submitted 2021-02-23; First posted 2021-02-26 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Arteriovenous Malformations
MeSH Terms: conditions — Arteriovenous Malformations | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — EDTA and DNA Streck blood tubes
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: blood sample — During the arteriography a peripheral venous sampling

SUMMARY:
Cerebral and medullary arteriovenous malformations (AVMs) lead to arterial and venous networks to communicate pathologically, creating an arteriovenous shunt. The occurrence of intracranial haemorrhage is the most important prognostic factor of AVMs because it is associated with a significant morbidity and mortality. The genetic, molecular and cellular mechanisms that cause vascular malformations of the central nervous system are partially known and the influence of genetic damage on the prognosis of AVMs is poorly known.

DETAILED DESCRIPTION:
Cerebral and medullary arteriovenous malformations (AVMs) are morphologically abnormal vessels located on the surface or in the cerebral or medullary parenchyma. These vascular lesions cause the arterial and venous networks to communicate pathologically, creating an arteriovenous shunt.

The prevalence of cerebral Cerebral and medullary AVMs in general population is difficult to establish given the rarity of the condition. However, it is estimated at around 1 per 10,000 inhabitants (0.01%). About 15-20% of the cerebral vascular accidents are asymptomatic at the time of diagnosis. The occurrence of intracranial haemorrhage is the most important prognostic factor because it is associated with a significant morbidity and mortality. The management of an AVM is usually carried out in a multidisciplinary way, combining interventional neuroradiology, neurosurgery and vascular neurology.

The genetic, molecular and cellular mechanisms that cause vascular malformations of the central nervous system are partially known. Several recent research works highlight mutations in the RAS-MAPK or MAPK-ERK signalling pathway in AVMs. In cases of cerebral AVMs considered to be sporadic, a somatic KRAS/BRAF mutation has recently been demonstrated in tissue samples of operated AVMs.

Except in the case of Hereditary Haemorrhagic Telangiectasia (HHT or Rendu-Osler-Weber syndrome), the influence of genetic damage on the prognosis of AVM is poorly known. It is also interesting to note that genetic screening is not routinely performed in patients with cerebro-medullary AVMs and that therefore the prevalence of these clinical entities in patients with AVMs is not known.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a vascular malformation of the cerebral or medullary identified on diagnostic imaging (angio-CT, angio-MRI or diagnostic angiography) for which clinical monitoring alone or intervention (endovascular treatment, surgery or radiosurgery) is planned in the centres participating in the research.

Exclusion Criteria:

* Pregnant, parturient or breastfeeding woman

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The recruited population will be index cases with cerebrovascular cerebral vascular malformations treated in the participating centres
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-02-17 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Genetic mutation | limit of 12 month
  Presence of a pathogenic mutation in one of the genes tested in the panel or identification of a pathogenic mutation following sequencing of the exome and/or transcriptome of the patient and/or his/her parents.

CONTACTS AND LOCATIONS:
Overall Officials: Stanislas Smajda, MD, Principal Investigator — Fondation Ophtalmologique Adolphe de Rothschild
Locations (1):
- HOPITAL FONDATION Adolphe de ROTHSCHILD, Paris, France